CLINICAL TRIAL: NCT02790125
Title: A Randomized, Double Blind Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986166 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IM018-001
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — BMS-986166

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Panel 1 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Single oral dose of solution as specified
  Interventions: Drug: BMS-986166; Drug: Placebo matching BMS-986166
- Dose Panel 2 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Single oral dose of solution as specified
  Interventions: Drug: BMS-986166; Drug: Placebo matching BMS-986166
- Dose Panel 3 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Single oral dose of solution as specified
  Interventions: Drug: BMS-986166; Drug: Placebo matching BMS-986166
- Dose Panel 4 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Multiple ascending solid dose formulation as specified
  Interventions: Drug: BMS-986166; Drug: Placebo matching BMS-986166
- Dose Panel 5a/b/c (Experimental): BMS-986166
  Single oral solid dose formulation under fasting/fed/fasting with famotidine conditions
  Interventions: Drug: BMS-986166

INTERVENTIONS:
Drug: BMS-986166
Drug: Placebo matching BMS-986166
  Arms: Dose Panel 1; Dose Panel 2; Dose Panel 3; Dose Panel 4

SUMMARY:
The primary purpose of this study is to determine if single doses of BMS-986166 are safe and well tolerated in healthy male subjects and female subjects of non-childbearing potential.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy female subjects of non-childbearing potential or male subjects as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations
* Ages 18 to 55 years
* Female subjects must provide documentation of an acceptable method of surgical sterilization or meet the protocol criteria for menopause

Exclusion Criteria:

* Any acute or chronic medical illness judged to be clinically significant by the Investigator and/or Sponsor medical monitor
* Any acute or chronic bacterial, fungal or viral infection, including tuberculosis, HIV, hepatitis B or hepatitis C, as defined in the protocol
* History of heart disease, neurological disease, eye disorders or gastrointestinal disorders or surgery (including cholecystectomy)
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs or clinical laboratory tests
* Smoking or nicotine use, drug or alcohol abuse within 6 months of starting the study

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-07-28 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of All Adverse Events (AEs) | Baseline Day -1 to Day 65
Incidence of Serious Adverse Events (SAEs) | Baseline Day -1 to Day 65
Severity of all All Adverse Events (AEs) | Baseline Day -1 to Day 65
Change from baseline in electrocardiogram(ECG) results | Baseline Day -1 to Day 35
Change from baseline in body temperature | Baseline Day -1 to Day 35
Change from baseline in respiratory rate | Baseline Day -1 to Day 35
Change from baseline in seated blood pressure | Baseline Day -1 to Day 35
Change from baseline in heart rate | Baseline Day -1 to Day 35
Change from baseline in clinical laboratory test results | Baseline Day -1 to Day 35
  Clinical laboratory testing to include Chemistry analytes and Hematology analytes.
Change from baseline in continuous cardiac monitoring data | Baseline Day -1 to Day 35
Change from baseline in physical examination findings | Baseline Day -1 to Day 35

SECONDARY OUTCOMES:
Mean difference in nadir heart rate (HR) and its time-matched HR on Day -1 | Day -1 to Day 4
Largest decrease in HR from time-matched Day -1 baseline | Day -1 to Day 4
Time to nadir HR from time 0 hour (predose) | Day -1 to Day 4
Percent reduction in HR at nadir from time-matched Day -1 HR value | Day -1 to Day 4
Mean change from baseline in HR values by timepoint for BMS-986166-treated versus placebo-treated subjects where the baseline is defined as time-matched Day -1 HR value | Day -1 to Day 7
Mean difference in absolute lymphocyte count (ALC) values and its time-matched ALC on Day -1 in BMS-986166- treated versus placebo-treated subjects | Day -1 to Day 4
Largest decrease in ALC from time-matched Day -1 baseline | Day -1 to Day 4
Time to nadir ALC from time 0 hour (predose) | Day -1 to Day 4
Percent reduction in ALC at nadir from time-matched Day -1 value | Day -1 to Day 4
Mean change from baseline in ALC values by timepoint for BMS-986166-treated versus placebo-treated subjects where the baseline is defined as time-matched Day -1 ALC value | Day -1 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LLC, Austin, Texas, United States

REFERENCES:
- [Derived] Singhal S, Girgis IG, Xie J, Dutta S, Shevell DE, Throup J. The safety and pharmacokinetics of a novel, selective S1P1R modulator in healthy participants. Expert Opin Investig Drugs. 2020 Apr;29(4):411-422. doi: 10.1080/13543784.2020.1742322. PMID 32306792
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx